CLINICAL TRIAL: NCT06871358
Title: The Effect of Pre- and Post-Administration of 80 mg Atorvastatin on Hs-CRP/Albumin Ratio in Reducing Thrombus Burden in STEMI Patients Undergoing Primary PCI
Brief Title: The Effect of Atorvastatin 80 mg on Hs-CRP/Albumin Ratio in Reducing Thrombus Burden in PCI-STEMI Patients
Acronym: PCI-STEMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Sebelas Maret (Other)
Responsible Party: Principal Investigator, Yos Akbar Irmansyah, Senior Cardiology Resident, Cardiology Department of Medical Faculty of Universitas Sebelas Maret, Universitas Sebelas Maret
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2.149/VIII/HREC/2024; RSUD Dr. Moewardi (Other: Universitas Sebelas Maret)
Record Dates: First submitted 2025-03-03; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: STEMI (STE-ACS); Primary PCI for STEMI
Keywords: Atorvastatin; hs-CRP; Albumin; TIMI Thrombus Grade; Thrombus Burden
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Atorvastatin

STUDY DESIGN:
Intervention Model Description: 40 STEMI patients undergoing primary PCI at Dr. Moewardi General Hospital participated in this experimental investigation. Using a double-blind technique, subjects were randomized into two groups: one receiving 80 mg of atorvastatin and the other's don't. Prior to and following primary PCI, levels of albumin and hs-CRP were assessed also their correlation with TIMI Thrombus Grade.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atorvastatin (Active Comparator): receiving 80 mg of atorvastatin in emergency department before primary PCI
  Interventions: Drug: Atorvastatin 80mg
- Placebo (Placebo Comparator): Did not receive Atorvastatin 80 mg before Primary PCI
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin 80mg — 80 mg of Atorvastatin are loading in first medical contact (Emergency Department) before primary PCI
  Other Names: Loading Atorvastatin 80 mg
  Arms: Atorvastatin
Drug: Placebo — Only given a loading DAPT without loading Atorvastatin 80 mg
  Arms: Placebo

SUMMARY:
40 STEMI patients who underwent primary PCI were subsequently allocated into two groups via a double-blind randomization method: An Atorvastatin 80 mg group and the control group.

Levels of hs-CRP and albumin were assessed for both groups upon presentation at the emergency department before to initial PCI and were re-evaluated 24 hours after primary PCI. Thrombus burden was assessed using angiography with the TIMI Thrombus grade.

DETAILED DESCRIPTION:
This study encompasses 40 STEMI patients who underwent primary PCI at Dr. Moewardi General Hospital in Central Java, Indonesia, between September and October. This study employed an experimental design with a pre-and-post technique, with participants recruited through sequential sampling. Patients were subsequently allocated into two groups via a double-blind randomization method. A treatment group was administered a loading dose of high-intensity statin (80 mg atorvastatin) upon initial presentation at the emergency department (ED), whereas the control group received no such intervention. Both cohorts received therapy in accordance with established guidelines prior to performing primary PCI.

Levels of hs-CRP and albumin were assessed for both groups upon presentation at the emergency department before to initial PCI. In the treatment group, a second 80 mg dose of atorvastatin was provided 24 hours after the original dose. Both hs-CRP and albumin levels were re-evaluated 24 hours after primary PCI in both the control and treatment cohorts.

Thrombus burden was assessed using angiography with the TIMI Thrombus grade

ELIGIBILITY:
Inclusion Criteria:

* STEMI with onset less than 24 hour and undergo a Primary PCI

Exclusion Criteria:

* STEMI beyond 24 hours from the onset of chest pain
* Prior statin therapy within the preceding 24 hours
* Hypersensitivity to statins, pregnancy, lactation, severe inflammatory conditions including active liver dysfunction, chronic kidney disease (eGFR <30 mL/min), autoimmune disorders, malignancy, severe malnutrition, and
* Contraindications to statin administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
hs-CRP/Albumin ratio | From enrollment to the end of treatment at 3 days
  The administration of 80 mg atorvastatin significantly reducing the hs-CRP/Albumin ratio (Δ 0.35 ± 0.67; p < 0.001) if compared to the control group

SECONDARY OUTCOMES:
TIMI Thrombus Burden | From enrollment to door to balloon time (Less than 24 hour onset)
  Using a TIMI Thrombus Burden that measure while performing PCI, we analyze that High burden thrombus was correlated with elevated of hs-CRP/Albumin ratio (r = 0.562; p = 0.012; r > 0.05; p < 0.05). So, by reducing Hs-CRP/Albumin Ratio, it appears also reducing the TIMI Thrombus burden.

CONTACTS AND LOCATIONS:
Locations (1):
- RSUD Dr Moewardi, Surakarta, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
To prevent similarity in primary Data

REFERENCES:
- [Background] Elserafy AS, Farag NM, El Desoky AI, Eletriby KA. Effect of high-intensity statin preloading on TIMI flow in patients presenting with ST-elevation myocardial infarction undergoing primary percutaneous coronary intervention. Egypt Heart J. 2020 Jul 10;72(1):40. doi: 10.1186/s43044-020-00074-0. PMID 32651772
- [Background] Wasyanto T, Yasa A, Murti B. The Effect of Colchicine Administration on HsCRP Level and Mean Platelet Volume in Patients with Miocard Acute Infark. Indonesian Journal of Medicine. 2018 Jan 1;3(3):162-7
- [Background] Duman H, Cinier G, Bakirci EM, Duman H, Simsek Z, Hamur H, Degirmenci H, Emlek N. Relationship Between C-Reactive Protein to Albumin Ratio and Thrombus Burden in Patients With Acute Coronary Syndrome. Clin Appl Thromb Hemost. 2019 Jan-Dec;25:1076029618824418. doi: 10.1177/1076029618824418. PMID 30808220
- [Background] Karabag Y, Cagdas M, Rencuzogullari I, Karakoyun S, Artac I, Ilis D, Yesin M, Cagdas OS, Altintas B, Burak C, Tanboga HI. Usefulness of The C-Reactive Protein/Albumin Ratio for Predicting No-Reflow in ST-elevation myocardial infarction treated with primary percutaneous coronary intervention. Eur J Clin Invest. 2018 Jun;48(6):e12928. doi: 10.1111/eci.12928. Epub 2018 Apr 17. PMID 29577260
- [Background] Acet H, Guzel T, Aslan B, Isik MA, Ertas F, Catalkaya S. Predictive Value of C-Reactive Protein to Albumin Ratio in ST-Segment Elevation Myocardial Infarction Patients Treated With Primary Percutaneous Coronary Intervention. Angiology. 2021 Mar;72(3):244-251. doi: 10.1177/0003319720963697. Epub 2020 Dec 29. PMID 33371718
- [Background] Wang H, Liu Z, Shao J, Lin L, Jiang M, Wang L, Lu X, Zhang H, Chen Y, Zhang R. Immune and Inflammation in Acute Coronary Syndrome: Molecular Mechanisms and Therapeutic Implications. J Immunol Res. 2020 Aug 18;2020:4904217. doi: 10.1155/2020/4904217. eCollection 2020. PMID 32908939
- [Background] Salari N, Morddarvanjoghi F, Abdolmaleki A, Rasoulpoor S, Khaleghi AA, Hezarkhani LA, Shohaimi S, Mohammadi M. The global prevalence of myocardial infarction: a systematic review and meta-analysis. BMC Cardiovasc Disord. 2023 Apr 22;23(1):206. doi: 10.1186/s12872-023-03231-w. PMID 37087452
- [Background] Kadappu P, Jonnagaddala J, Liaw ST, Cochran BJ, Rye KA, Ong KL. Statin Prescription Patterns and Associations with Subclinical Inflammation. Medicina (Kaunas). 2022 Aug 14;58(8):1096. doi: 10.3390/medicina58081096. PMID 36013563
- [Background] Waksman R, Merdler I, Case BC, Waksman O, Porto I. Targeting inflammation in atherosclerosis: overview, strategy and directions. EuroIntervention. 2024 Jan 1;20(1):32-44. doi: 10.4244/EIJ-D-23-00606. PMID 38165117